CLINICAL TRIAL: NCT06314620
Title: Safety And Efficacy Of 8 Hourly Normal Saline Flushing With And Without Heparin Lock In Maintaining Small Bore Intercostal Chest Catheter (ICC) Patency ; A Prospective Pilot Study
Brief Title: Normal Saline Flushing With And Without Heparin Lock In Maintaining Small Bore Intercostal Chest Catheter (ICC) Patency
Acronym: SENSHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FF-2024-043
Record Dates: First submitted 2024-02-18; First posted 2024-03-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants who underwent ICC with normal saline flushing and heparin lock (Active Comparator): Participants who underwent intercostal chest catheter with normal saline flushing with heparin lock. Instillation done with 20 mls of Normal Saline flush followed by heparin saline lock, every 6 hours by a three way stopcock.
  Interventions: Drug: Heparin saline lock
- Participants who underwent ICC with normal saline flushing without heparin lock (Active Comparator): Participants who underwent intercostal chest catheter with normal saline flushing without heparin lock. Instillation done with 20 mls of Normal Saline flush , every 6 hours by a three way stopcock.
  Interventions: Other: Without heparin saline lock

INTERVENTIONS:
Drug: Heparin saline lock — Participants with intercostal chest catheter who underwent normal saline flushing with heparin saline lock
  Arms: Participants who underwent ICC with normal saline flushing and heparin lock
Other: Without heparin saline lock — Participants with intercostal chest catheter who underwent normal saline flushing without heparin saline lock
  Arms: Participants who underwent ICC with normal saline flushing without heparin lock

SUMMARY:
Pleural diseases are among the most common clinical problems encountered in healthcare settings in Malaysia and even worldwide. Most patients presented in a hospital setting with pleural diseases will need pleural aspirations or thoracentesis and chest drains for a variety of reasons. Healthcare providers will often be exposed to patients requiring pleural drainage hence it is important to be aware of safe techniques and procedures of insertion and also maintaining the pleural drainage systems to yield beneficial results.

Most often, smaller catheters were deemed to be less effective in view of slower drainage rates and associated with high risk of blockage. However presently , in tertiary hospital settings small bore intercostal chest catheters (SBICC) have become an alternative to large bore intercostal catheters (LBICC). SBICC has been found to be equally effective, less painful and easily tolerated by patients. Hence, proper maintenance of SBICC should be undertaken to reduce rates of occlusion and to yield most benefits from the pleural aspirations procedures.

British Thoracic Society in their latest guidelines recommends the use of small bore intercostal chest drain as the first choice in draining pleural effusions.

The success of draining pleural effusions with a SBICC has shown variable rates of success among different studies conducted. Most common issues faced are drain blockage and drain dislodgement.

There is limited data comparing the use of normal saline flushing versus fibrinolytic drug lock in maintaining patency of small bore intercostal chest drains in draining pleural effusions. This has lead us in conducting this research to compare the rates of partial or complete occlusions among normal saline flush with and without heparin saline lock in maintaining the patency of small bore intercostal chest catheter among patients with pleural diseases in Hospital Canselor Tuanku Muhriz, UKM requiring chest drains insertion.

DETAILED DESCRIPTION:
Hypothesis

1. Rate of occlusion is less in group with Heparin Saline lock.
2. Rate of occlusions is higher in patients with exudative effusions. e.g : Empyema, raised pleural fluid LDH, low pleural pH, positive pleural cultures.
3. Onset of ICC occlusions is lower in group with Heparin Saline lock.
4. There is no difference in blood parameters between 2 groups.
5. There are no apparent adverse effects between 2 groups.
6. Patients in group with Heparin Saline lock have lower numbers of fenestration occluded.

Significance of Research Pleural diseases are among the most common diseases encountered in tertiary hospitals in Malaysia. Healthcare providers will need to provide adequate drainage of pleural fluids to improve the treatment outcome of patients. One of the mainstays of treatment is to ensure adequate drainage by reducing the rate of blockage of chest drains. This study is a pilot study to determine the efficacy as well as to ascertain the safety profile of using normal saline vs heparin saline lock for small bore intercostal catheters among pleural disease patients.

Type of Study Study on the Safety and Efficacy of 8 Hourly Flushing of ICC with and without Heparin Saline Lock in Maintaining Patency of ICC (SENSHIP Trial) is a prospective open label randomized controlled trial , a pilot study of patients admitted with pleural diseases in need of small bore intercostal catheters in Hospital Canselor Tuanku Muhriz, HUKM.

Standard Of Care Current Standard of Care in managing ICC in pleural diseases follows the recommendation of British Thoracic Society Guidelines where it suggests for regular flushing of ICC. The guideline recommends flushing of the tube by instilling 20-30ml of Normal Saline flush every 6 to 8 hours by a three way stopcock. However, this guideline only recommends regular flushing with Normal Saline and no research has been conducted to compare the outcome of effusions drainage and rates of blockage in small bore chest tubes with different techniques of flushing. Despite regular flushing with Normal Saline solutions as recommended, the rate of blockages in ICC still remains high. Hence, by adapting the concept of Heparin Saline Lock in IJC to maintain the patency of the tubing, we would like to study the difference of regular 8 hourly Normal Saline flushing with and without Heparin Saline Lock in maintaining ICC. Participants in this study who are chosen into Heparin Saline Lock arm will be receiving approximately 2ml of Heparin Saline as locking solution in attempt to maintain the ICC tube.

This study will be conducted in all medical wards of Hospital Canselor Tuanku Muhriz, HUKM.

Sampling Population

This study will be conducted among inpatients in medical wards with pleural effusions requiring small bore intercostal chest catheters who had been screened and consented to be involved in this study. All participants will be randomly allocated into 2 groups :

1. Group without Heparin Saline Lock
2. Group with Heparin Saline Lock

The group with heparin saline lock will receive approximately 1-2mls Heparin Saline as a locking solution (depending on the length of catheter). The amount of Heparin Saline lock to be instilled will depends on the estimated catheter volume. After flushing, the catheter will be clamped for 1 hour and then unclamped after 1 hour. Data will then be collected from 2 different groups to be analysed.

Sample Size Sample size is calculated using 'Select Statistical Online Calculator'; using 2 sample comparisons of percentages. There were no previous study comparing the efficacy and safety of Heparin Saline Lock vs Normal Saline Lock in maintaining the patency of small-bore ICC, thus the sample size calculated using the study conducted previous study by Claire. The study reported a 32% reduction in pleural fluid volume on CT over 3 days in the irrigation group compared to a 15% reduction in patients treated with chest-tube drainage alone (p<0.04).

Estimated sample size for two-sample comparison of percentages

Assumptions:

Alpha = 5% (two-sided) Power = 80% Intervention (Heparin) = 32% Standard (NS) = 15%

Estimated sample size:

n1 (Heparin) = 96 n2 (NS) = 96

Missing data estimated to be 10%, therefore minimum total sample required is 212 (Intervention = 106 , Standard = 106)

However, as this is a pilot study, the estimated sample size taken for this study is 20% from the calculated sample size with missing data estimated to be 10%.

Estimated sample size :

n1 (Heparin) : 20 n2 (NS) : 20

Therefore, minimum total sample needed is 40

Statistical Analysis

Statistical analyses will be performed with SPSS v23 software. Descriptive statistics, such as the frequency (n), arithmetic mean (x), and standard deviation (SD), are presented for normally distributed variables. A 2- sample independent test for mean and proportions will be used to calculate the statistical significance value between the 2 independent groups. Statistical significance was defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

• All patients admitted in medical wards for pleural effusion who had small bore intercostal catheters inserted.

Exclusion Criteria:

* Patients with hydropneumothorax with small bore intercostal catheters
* Patients with septated effusion planned for intrapleural fibrinolysis
* Patients with severe coagulopathy

  * INR ≥ 1.5
  * PT > 37s
  * aPTT > 100s
* Patients with thrombocytopenia of less than 50 x 109/L
* Patients who has not consented to be involved in the study
* Patients with indwelling pleural catheters
* Unconscious patients will be excluded from this study
* Patients with poor GCS score will be excluded from this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
To compare the rate (in percentage) of occlusions of intercostal chest catheter in participants underwent normal saline flushing with and without heparin lock | From the time of randomization to the time of the end of study up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.

SECONDARY OUTCOMES:
To determine the onset of intercostal chest catheter occlusions (in hours) | From the time of randomization to the time of the end of study up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.
To determine the change of hemoglobin (in g/dL) post ICC insertion | From the time of randomization to the time of the end of study up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.
To determine the change of platelet (in 10 9/L) post ICC insertion | From the time of randomization to the time of the end of study up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.
To determine the adverse effects of heparin saline lock | From the time of randomization to the time of the end of study up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.
To assess the number of fenestrations occluded (in numbers from 0-5) with fibrin or blood clots | From the time of randomization to the time of the end of study up to up to 30 days post insertion of chest drain
  Participants who underwent intercostal chest catheter insertion who received normal saline flushing with and without heparin lock.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS (IIUM), Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Horsley A, Jones L, White J, Henry M. Efficacy and complications of small-bore, wire-guided chest drains. Chest. 2006 Dec;130(6):1857-63. doi: 10.1378/chest.130.6.1857. PMID 17167009
- [Result] Maskell N; British Thoracic Society Pleural Disease Guideline Group. British Thoracic Society Pleural Disease Guidelines--2010 update. Thorax. 2010 Aug;65(8):667-9. doi: 10.1136/thx.2010.140236. No abstract available. PMID 20685739
- [Result] Keeling AN, Leong S, Logan PM, Lee MJ. Empyema and effusion: outcome of image-guided small-bore catheter drainage. Cardiovasc Intervent Radiol. 2008 Jan-Feb;31(1):135-41. doi: 10.1007/s00270-007-9197-0. Epub 2007 Oct 18. PMID 17943347
- [Result] Davies HE, Merchant S, McGown A. A study of the complications of small bore 'Seldinger' intercostal chest drains. Respirology. 2008 Jun;13(4):603-7. doi: 10.1111/j.1440-1843.2008.01296.x. Epub 2008 Apr 14. PMID 18422864
- [Result] Porcel JM, Azzopardi M, Koegelenberg CF, Maldonado F, Rahman NM, Lee YC. The diagnosis of pleural effusions. Expert Rev Respir Med. 2015;9(6):801-15. doi: 10.1586/17476348.2015.1098535. Epub 2015 Oct 8. PMID 26449328
- [Result] Parulekar W, Di Primio G, Matzinger F, Dennie C, Bociek G. Use of small-bore vs large-bore chest tubes for treatment of malignant pleural effusions. Chest. 2001 Jul;120(1):19-25. doi: 10.1378/chest.120.1.19. PMID 11451810
- [Result] Mehra S, Heraganahally S, Sajkov D, Morton S, Bowden J. The effectiveness of small-bore intercostal catheters versus large-bore chest tubes in the management of pleural disease with the systematic review of literature. Lung India. 2020 May-Jun;37(3):198-203. doi: 10.4103/lungindia.lungindia_229_19. PMID 32367840
- [Result] Collop NA, Kim S, Sahn SA. Analysis of tube thoracostomy performed by pulmonologists at a teaching hospital. Chest. 1997 Sep;112(3):709-13. doi: 10.1378/chest.112.3.709. PMID 9315804
- [Result] Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, Medford AR, Harvey JE, Darby M, Zahan-Evans N, Maskell NA. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J. 2015 Aug;46(2):456-63. doi: 10.1183/09031936.00147214. Epub 2015 May 28. PMID 26022948
- [Result] Goossens GA. Flushing and Locking of Venous Catheters: Available Evidence and Evidence Deficit. Nurs Res Pract. 2015;2015:985686. doi: 10.1155/2015/985686. Epub 2015 May 14. PMID 26075094
- [Result] Shaikh N. Heparin-induced thrombocytopenia. J Emerg Trauma Shock. 2011 Jan;4(1):97-102. doi: 10.4103/0974-2700.76843. PMID 21633576

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT06314620/Prot_SAP_ICF_000.pdf